CLINICAL TRIAL: NCT02858635
Title: Molecular Genetics of Suicidal Behavior: Study of Association Between Aggressive Impulsiveness and Genes of the Serotoninergic System
Brief Title: Molecular Genetics of Suicidal Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Créteil Hospital (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 7653
Record Dates: First submitted 2016-07-18; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Suicidal Behaviour
Keywords: Suicidal behaviour; Impulsivity; Genetics; Serotonin
MeSH Terms: conditions — Impulsive Behavior | interventions — Neuropsychological Tests; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Suicide attempters (Experimental): Clinical and neuropsychological assessment. Blood and saliva samples in order to answer objectives study.
  Interventions: Other: Clinical and neuropsychological assessment, Blood and saliva samples

INTERVENTIONS:
Other: Clinical and neuropsychological assessment, Blood and saliva samples — Clinical and neuropsychological assessment: impulsivity, aggressiveness, psychological pain, angor with specific scales and smartphone.

SUMMARY:
Suicide is a major health problem that causes annually a million death worldwide. In the stress-vulnerability model, suicidal behavior (SB) results from the interaction between an individual's predisposition and stressful condition. According to this model, individuals who carry a suicidal act when subjected to stress factors (environmental stress, depression, substance ...) are those which have a specific vulnerability.These vulnerabilities can be considered as clinical parameters (propensity to despair, aggressive and/or impulsive traits), neurobiological parameters (dysfunction of the serotonergic system, ...) and cognitive parameters (taking disadvantageous decision ...). Suicidal vulnerability is partly underpinned by genetic factors. The interest of current researches is to identify biomarkers that will improve the opportunities for early identification of subject with a risk for SB.

The four goals of this project are in the continuity of previous works team:

1. To determine whether combinations of the main serotonin-related genes may better contribute to the vulnerability to SB, than when they are considered independently.
2. To assess whether the associations between these genes and SB are modulated by childhood trauma, life events and stress response associated with these environmental factors.
3. To test the value of combined clinical, neuropsychological and genetic factor for suicide prevention, in a prospective study, in particularity impulsivity and gene gene interaction.
4. To investigate the association between events in real life (using ecological momentary assessment) and emotional response and suicidal ideation.

The investigators propose to use a multidisciplinary approach to answer these questions and, hence, be able to identify new prevention strategies for SB.

DETAILED DESCRIPTION:
Transversal study:

1500 patients with a personal history of suicide attempt will be recruited. Clinical, biological and neuropsychological assessments will be performed. The first objective of the study is to replicate the results already obtained regarding the association between serotonergic system genes and suicidal behaviour. The allele frequencies for different markers tested in suicidal and in control subjects with no history of suicidal behaviour will be compared. The patients that will be recruited will be compared to the control population already recruited for another project.

Prospective study: 554 patients hospitalized for a suicide attempt will will be evaluated, each 6 month, during the 2-years period of the study. Clinical, biological and neuropsychological assessments will be performed.

At the end of the inclusion visit, 60 participants will be assessed using ecological momentary assessment(ESM). They will be instructed to carry a smartphone with them for one week, and to record at each alarm signal daily life events, negative emotions, psychological pain, suicidal ideas, and specific attributions to these events. Participants will be signalled five times a day during the period. Subjects will be contacted by telephone halfway through the assessment period to monitor and encourage compliance.

ELIGIBILITY:
Inclusion Criteria:

* personal history of suicide attempt
* French Caucasian Western Europe and specifically have all four grandparents from a country in Western Europe (for genetics purposes)
* able to understand nature, aims, and methodology oh the study
* do not emphasize to leave during the time-study.

Exclusion Criteria:

* Pregnancy
* Not able to speak, read and understand French
* Patient on protective measures (guardianship or trusteeship)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1982 (Actual)
Dates: Start 2001-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
occurrence of suicide attempt | up to 6 months
  occurrence of a suicide attempt will be assessed by the Columbia History Form at each visit

SECONDARY OUTCOMES:
suicidal ideation | up to 7 days
  suicidal ideation will be assessed by scale for suicidal ideation (SSI) self-assessments (with a smartphone) by Likert scales, 5 times per day during 7 days.
number of suicide attempt | 1 hour
  assessed by clinical interview
type of suicide attempt | 1 hour
  assessed by clinical interview
lethality of suicide attempt | 1 hour
  assessed by Risk-Rescue Rating Scale (RRRS)
anger | 1 hour
  assessed by State-Trait Anger Expression Inventory (STAXI scale)
Impulsivity | 1 hour
  assessed by barratt impulsiveness scale (BIS scale)
aggressiveness | 1 hour
  assessed by buss durkee hostility inventory (BDHI)
psychological pain | 1 hour
  assessed by Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided